CLINICAL TRIAL: NCT04942678
Title: The Impact of Therapy Dogs on Anxiety and Emotional Management in the Pediatric Emergency Department
Status: Completed | Type: Observational
Sponsor: University of Louisville (Other)
Responsible Party: Principal Investigator, Michelle D. Stevenson, Professor of Pediatrics Director of Research Development, Department of Pediatrics, University of Louisville Norton Children's Medical Group, Affiliated with the U of L School of Medicine, University of Louisville
Other Study IDs: 21.0190
Record Dates: First submitted 2021-03-25; First posted 2021-06-28 (Actual); Last update posted 2022-03-17 (Actual); Status verified 2022-03

CONDITIONS: Anxiety; Emotional Regulation
Keywords: Pediatric Emergency Medicine; Therapy Animals; Animal Assisted Therapy; Anxiety; Emotional Regulation
MeSH Terms: conditions — Anxiety Disorders; Emotional Regulation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pediatric patients ages 4-7 years old in the Pediatric Emergency Department: Patients will receive a 10-minute visit with therapy dog and child life handler
  Interventions: Behavioral: 10-minute visit with therapy dog and child life specialist handler
- Pediatric patients ages 8-12 years old in the Pediatric Emergency Department: Patients will receive a 10-minute visit with therapy dog and child life handler
  Interventions: Behavioral: 10-minute visit with therapy dog and child life specialist handler

INTERVENTIONS:
Behavioral: 10-minute visit with therapy dog and child life specialist handler — A visit from a therapy dog and child life specialist will occur which will last for approximately 10 minutes. Parents and patients will be asked to sanitize their hand prior to the visit. The child life specialist will be instructed to have ad lib conversation with the family. The dog will remain on a leash during the visit. The patient will be free to pet the therapy dog if they wish.

SUMMARY:
The purpose of this study is to assess the impact of therapy dogs on children's anxiety and emotional management during a visit to the pediatric emergency department.

ELIGIBILITY:
Inclusion Criteria:

* Children with a SUD score of 30 or higher indicated by the caregiver

Exclusion Criteria:

* Active infection: abscesses, fever, respiratory issues, vomiting
* Patients presenting for burn care, dog bite, ESI triage category 1 or 2, or transferred from outside facilities
* Sterile procedures
* Oncology patients / patients with known neutropenia in past medical history
* Parent/caregiver or patient fear of dogs
* Parent/caregiver or patient allergy to dogs
* Dog bite injury
* Already underwent procedure during their visit

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Patients will be recruited at both Norton Children's Hospital Emergency Department and Norton Children's Medical Center Emergency department.
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2021-05-25 (Actual); Primary Completion 2021-07-26 (Actual); Study Completion 2021-07-26 (Actual)

PRIMARY OUTCOMES:
Change in observed anxiety score as measured by Child Emotional Manifestation Scale (CEMS) before and after therapy dog visit | change from baseline at 20 minutes after intervention
  To determine the change in emotional management in children aged 4-12 years after a visit from a therapy dog and child life specialist handler, as measured by an observed CEMS score (Children's Emotional Management Scale) before and after the visit. This will be completed by an investigator. Scores range from 5-25, with higher scores indicating higher levels of observed anxiety.

SECONDARY OUTCOMES:
Change in perceived anxiety level of patient by parent as measured by Subjective Units of Distress Scale (SUDs) before and after therapy Dog Visit | change from baseline at 20 minutes after intervention
  To determine the change in perceived level of child anxiety as reported by parents after a visit with a therapy dog and child life specialist handler. This will be measured using the Subjective Unit of Distress (SUD) score. Scores range from 0-100 with higher scores indicating higher levels of perceived anxiety by the parent.
Overall Parent Satisfaction | Immediately after completion of intervention
  Parents will complete a survey describing their satisfaction with their visit

CONTACTS AND LOCATIONS:
Overall Officials: Michelle D Stevenson, MD, MS, Principal Investigator — University of Louisville
Locations (1):
- Norton Children's Hospital, Louisville, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No